CLINICAL TRIAL: NCT04771247
Title: Endoscopic Cardiac Band Ligation (CLEAR) Without Sleeve Stenosis for the Management of Refractory GERD After Laparoscopic Sleeve Gastrectomy (LSG)
Brief Title: Endoscopic Cardiac Band Ligation for the Management of Refractory GERD After Laparoscopic Sleeve Gastrectomy
Acronym: CLEAR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB approval withheld
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00277820
Record Dates: First submitted 2021-02-23; First posted 2021-02-25 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: GERD; Bariatric Surgery; Laparoscopic Sleeve Gastrectomy
Keywords: CLEAR; Antireflux procedure; LSG; GERD
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: Prospective, single center, pilot clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CLEAR (Experimental): Patients with GERD post LSG will undergo CLEAR (cardia band ligation).
  Interventions: Procedure: Cardia Band Ligation

INTERVENTIONS:
Procedure: Cardia Band Ligation — Patients will undergo cardia band ligation at the level of the GEJ.

SUMMARY:
GERD is a prevalent condition worldwide, estimated to be around 20-30 % in North America. Obesity is rapidly increasing with an estimated prevalence of 66% in the adult population in the United States. Presently, bariatric interventions are the only sustainable method to address morbid obesity and its resulting comorbidities. One of the most common restrictive surgeries includes laparoscopic sleeve gastrectomy (LSG). Although very effective for treating obesity, some of these surgeries might cause deleterious effects regarding GERD, due to anatomical modifications. Refractory GERD is defined by lack of symptom control on maximum dose of PPI therapy. Cardia Band Ligation Anti-reflux (CLEAR) procedure utilizes multiple band ligations at the cardia in a 270-degree fashion, resulting in tissue necrosis and scar formation, narrowing the GE junction and enhancing the flap valve system. The investigators hypothesized that CLEAR can be a safe and efficient intervention to improve post bariatric GERD.

DETAILED DESCRIPTION:
GERD is a prevalent condition worldwide, estimated to be around 20-30 % in North America. Obesity is rapidly increasing with an estimated prevalence of 66% in the adult population in the United States. GERD symptoms are common in the obese population with data showing weekly GERD symptoms in 34.6% and erosive esophagitis 26.9% in people with BMI > 30 Kg/m^2. Reflux is associated with complications such as esophagitis, Barrett's Esophagus and ultimately esophageal adenocarcinoma. Presently, bariatric interventions are the only sustainable method to address morbid obesity and its resulting comorbidities. There are endoscopic and surgical bariatric interventions. Bariatric surgery has been shown to be an effective and efficient means of achieving significant weight loss in obese individuals. One of the most common restrictive surgeries includes laparoscopic sleeve gastrectomy (LSG). Although very effective for treating obesity, some of these surgeries might cause deleterious effects regarding GERD, due to anatomical modifications. LSG can increase the incidence of GERD, which may be explained from the changes in the angle of His and by increasing intragastric pressure. Pharmacological therapy with proton pump inhibitors (PPI), H2 blockers and lifestyle changes are first line forms of treatment utilized to control the symptoms related to GERD. However, patients who use pharmacological treatment experience reduction in quality of life and seek alternative options. Refractory GERD is defined by lack of symptom control on maximum dose of PPI therapy. Moreover, due to the anatomical changes associated with bariatric surgeries, the traditional surgical and endoscopic techniques (TIF, Nissen Fundoplication) used to treat GERD in the general population are not suitable for these patients. With the current trend of an increase of bariatric surgery and thus GERD that arises after these surgeries, new innovative techniques to treat GERD are needed, especially in PPI averse or non-responsive patients. Cardia Band Ligation Anti-reflux (CLEAR) procedure utilizes multiple band ligations at the cardia in a 270-degree fashion, resulting in tissue necrosis and scar formation, narrowing the GE junction and enhancing the flap valve system. The investigators will perform CLEAR by placing 4 bands at the GEJ. The investigators hypothesized that CLEAR can be a safe and efficient intervention to improve post bariatric GERD.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients who underwent surgical bariatric weight loss procedures with post-surgical GERD (LSG), not responding to once daily PPI therapy.
* Obese patients who underwent surgical bariatric weight loss procedures with post-surgical GERD (LSG) who respond to maximum therapy with PPI + H2 blocker but are PPI averse or who refuse surgical therapy (conversion to RYGBP).
* Patients older than 18 years and younger than 75 years of age at time of consent.
* Patients able to provide written informed consent on the IRB/EC-approved informed consent form
* Patients willing and able to comply with study requirements for follow-up

Exclusion Criteria:

* Any patient with no prior surgical bariatric intervention.
* Pre-existing esophageal stenosis/stricture preventing advancement of an endoscope during screening/baseline EGD.
* Esophageal, gastric or duodenal malignancy.
* Severe medical comorbidities precluding endoscopy, or limiting life expectancy to less than 2 years in the judgment of the endoscopist.
* Uncontrolled coagulopathy or inability to be off anticoagulation or anti-platelet medication (ASA, Plavix) for 1 week prior to and 2 weeks after each endoscopy
* Active fungal esophagitis, Grade C or D esophagitis.
* Hiatal hernias > 2 cm or para-esophageal hernias.
* Known portal hypertension, visible esophageal or gastric varices, or history of esophageal varices.
* General poor health, multiple co-morbidities placing the patient at risk, or otherwise unsuitable for trial participation.
* Pregnant or planning to become pregnant during period of study participation.
* Patient refuses or is unable to provide written informed consent.
* Prior surgical or endoscopic anti-reflux procedure.
* Persistent dysphagia score greater than 0.
* Vomiting more than once a week.
* Biopsy-proven Barrett's esophagus.
* HREM showing marked ineffective esophageal motility (defined by ≥ 5 weak or failed swallows per Chicago Classification v 3.0), esophagogastric outflow obstruction (EGJOO) or achalasia.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Change in GERD-HQRL/RSI score | Baseline and 6 months
  Change in symptoms assessed by GERD-HQRL/RSI score at 6 months.
Change in pH monitoring | Baseline and 6 months
  Change in objective pH monitoring at 6 months.

SECONDARY OUTCOMES:
Mean change on the percentage of acid exposure time (% AET) | Baseline and 6 months
  Changes in acid exposure time from baseline.
Safety of CLEAR procedure as assessed by treatment-related adverse events | Up to 6 months
  Assess overall safety (treatment-related adverse events) of CLEAR procedure defined by the ASGE-Lexicon classification.
Rate of dysphagia post CLEAR | 6-12 months
  Percentage of patients who develop dysphagia of any grade, associated with esophageal or gastric cardia stricture requiring dilation after CLEAR procedure.
PPI discontinuation | 6 months
  Percentage of patients who no longer require PPI at 6 months post CLEAR.
PPI discontinuation | 12 months
  Percentage of patients who no longer require PPI at 12 months post CLEAR.
Treatment failure | 6 months
  Defined as less than 50% improvement in GERD HQRL/RSI score or pH monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Olaya I Brewer Gutierrez, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Seleem WM, Hanafy AS, Mohamed SI. Endoscopic management of refractory gastroesophageal reflux disease. Scand J Gastroenterol. 2018 Apr;53(4):390-397. doi: 10.1080/00365521.2018.1445775. Epub 2018 Feb 28. PMID 29488430